CLINICAL TRIAL: NCT05370443
Title: Effectiveness of an Online Life Skills-based Intervention on Depression, Anxiety and Stress Among Arabic Adolescents in Klang Valley, Malaysia: Protocol for a Cluster-randomized Controlled Trial
Brief Title: Effectiveness of an Online Life Skills-based Intervention on Mental Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, YOSRA MOHAMED M SHERIF, Principal Investigator, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JKEUPM-2021-912
Record Dates: First submitted 2022-05-06; First posted 2022-05-11 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Mental Disorder in Adolescence
Keywords: Depression, Anxiety Stress, Life Skills, Arabic adolescents
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: This study is quantitative in nature and experimental in design. Specifically, this is a parallel cluster-randomized controlled trial. The schools will be the unit of randomisation (clusters). Arabic schools will be randomised in a 1:1 ratio to be either in the intervention (Life Skills educational program) or control group (waiting list). The participants will be asked to fill out the online form of the DASS-21 questionnaires (the screening stage). Then participants with a score of mild to extra-sever on at least one (depression, stress or anxiety) will be included in the life skills intervention study and will fill the second two parts of the questionnaires (GES and Brief Cope Scale).
Who Masked: Participant, Outcomes Assessor
Masking Description: No one in the control groups will know what the experimental groups will be offered. The the statistician who will perform the primary analyses will be blinded to group allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Life Skills intervention group (Experimental): The participants in the intervention group will receive eight sessions of the online life skills educational program via the zoom platform for eight weeks. Each session will last for 1-hour. All the participants will receive a short reminder SMS for enrolling in the online session. The assessment for all students will be done at baseline, immediate and 3-months post-intervention.
  Interventions: Behavioral: Life Skills education program
- control group (No Intervention): Participants in the control group will receive no intervention during the study period. However, they will receive the same educational activities after finishing study. They will answer the same questionnaires at baseline, immediately following the intervention, and three months later.

INTERVENTIONS:
Behavioral: Life Skills education program — The World Health Organization (WHO), describes life skills as "abilities for adaptive and positive behaviour that enables individuals to deal effectively with the demands and challenges of everyday life". Life Skills Education includes activities that support critical and creative thinking, coping with emotions and stress, self-awareness and empathy, decision-making and problem-solving, communication skills, and interpersonal relations.
  Arms: Life Skills intervention group

SUMMARY:
It is a parallel cluster randomised controlled trial designed to assess the effectiveness of an online life skills education in reducing depression, anxiety, and stress and improving self-efficacy and coping skills among Arabic secondary school students at Arabic schools in Klang Valley in Malaysia.

DETAILED DESCRIPTION:
Children and adolescents' mental health is a global public health issue. Worldwide, it is estimated between 10% and 20% of children and adolescents suffer from mental health problems. Depression and anxiety are the most frequently encountered mental disorders which significantly impact children and adolescents. These disorders have been shown to increase the risk of adverse outcomes such as impairment, loss of productivity and community involvement, decreased educational performance, increased likelihood of engaging in risky behaviours, disability, and increased self-harm and suicide rates. Migrant children and adolescents are at increased risk of these mental disorders, mainly Arabic immigrants. Arab adolescents face additional challenges such as high illiteracy rates, inadequate health services and poor access to health facilities, especially mental health facilities. There is also a clear trend of the increasing burden of mental disorders in the Arabic countries from 1990 to 2015 compared to the global average. This study examines the effectiveness of an online life skills-based intervention in reducing depression, anxiety and stress and improving self-efficacy and coping skills among Arabic secondary school students in Klang Valley in Malaysia. The life skills intervention modules and activities will be developed based on the WHO and UNICEF guidelines for implementing life skills. This program will also undergo a process of consultations with a group of experts. The intervention group will receive education videos and discussion sessions that will target self-awareness, Empathy, Interpersonal relationship skills, Communication skills, Critical and creative thinking, problem-solving, decision-making, and coping with stress and emotion. The sessions will be carried out per week for 1 hour for eight consecutive weeks via the zoom platform. Before conducting the intervention, all the participants will receive a short reminder SMS for enrolling in the online session. The control group will receive the education program after finishing the study.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for schools are:

  * Arabic schools that agree to participate.
  * The Arabic schools are located in Klang Valley.

The inclusion criteria for students:

* Arabic Students aged from 14 to 18 years old.
* students who give the assent and consent from their parents.
* Students who have scored mild to extremely severe score in depression, anxiety and stress based on baseline assessment (screening stage).

Exclusion Criteria:

* The exclusion criteria for schools are:

  * non-Arabic schools that have Arabic students.
  * Schools that refuse to participate in the study.

The exclusion criteria for students:

* students who refuse to participate.
* Students who have hearing limitations because they cannot interact during the online session.
* Students who have been diagnosed or treated for mental health problems before based on their school file because it may interfere with the effect of the program.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 339 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Change in the depression, anxiety and stress mean scores | Measurement will be pre-intervention(baseline), immediately post-intervention and 3 months post-intervention
  Depression, Anxiety Stress Scales-21 ( DASS-21). The DASS-21 is a set of three self-report scales designed to measure depression, anxiety, and stress. Each of the three sets of the DASS21 scales include seven items with a 4-point Likert scale. The minimum and maximum DASS21 scores are 0 and 21 for each subscale. Higher scores indicate higher levels of problems.

SECONDARY OUTCOMES:
Change in the Self-efficacy mean score | Measurement will be pre-intervention(baseline), immediately post-intervention and 3 months post-intervention
  The General Self-Efficacy Scale (GES). The GES is a 10-item psychometric scale rated on a 4-point Likert scale, ranging from 10-40, and a higher score indicates more self-efficacy. It is used to assess the strength of an individual's belief in his or her own ability to respond to new situations, obstacles, or life stresses.
Change in coping skills mean score | Measurement will be pre-intervention(baseline), immediately post-intervention and 3 months post-intervention
  Brief COPE Inventory is a self-report questionnaire consisting of 28 statements with a 4-point Likert scale to evaluate 14 different ways of coping with stressful situations. The minimum and maximum scores on the original Brief COPE questionnaire are 2 and 8, respectively, for each subscale. Higher scores reflect a higher tendency to implement the corresponding coping strategies

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Z Fattah Azman, Study Chair — UPM
Locations (1):
- Arabic schools in Klang Valley, Malaysia, Serdang, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mohammadzadeh M, Awang H, Ismail S, Kadir Shahar H. Improving emotional health and self-esteem of Malaysian adolescents living in orphanages through Life Skills Education program: A multi-centre randomized control trial. PLoS One. 2019 Dec 26;14(12):e0226333. doi: 10.1371/journal.pone.0226333. eCollection 2019. PMID 31877163
- [Result] van Loon AWG, Creemers HE, Beumer WY, Okorn A, Vogelaar S, Saab N, Miers AC, Westenberg PM, Asscher JJ. Can Schools Reduce Adolescent Psychological Stress? A Multilevel Meta-Analysis of the Effectiveness of School-Based Intervention Programs. J Youth Adolesc. 2020 Jun;49(6):1127-1145. doi: 10.1007/s10964-020-01201-5. Epub 2020 Feb 7. PMID 32034632
- [Result] Jamali S, Sabokdast S, Sharif Nia H, Goudarzian AH, Beik S, Allen KA. The Effect of Life Skills Training on Mental Health of Iranian Middle School Students: A Preliminary Study. Iran J Psychiatry. 2016 Oct;11(4):269-272. PMID 28050189
- [Result] Singla DR, Waqas A, Hamdani SU, Suleman N, Zafar SW, Zill-E-Huma, Saeed K, Servili C, Rahman A. Implementation and effectiveness of adolescent life skills programs in low- and middle-income countries: A critical review and meta-analysis. Behav Res Ther. 2020 Jul;130:103402. doi: 10.1016/j.brat.2019.04.010. Epub 2019 Apr 26. PMID 31146889
- [Result] Charara R, Forouzanfar M, Naghavi M, Moradi-Lakeh M, Afshin A, Vos T, Daoud F, Wang H, El Bcheraoui C, Khalil I, Hamadeh RR, Khosravi A, Rahimi-Movaghar V, Khader Y, Al-Hamad N, Makhlouf Obermeyer C, Rafay A, Asghar R, Rana SM, Shaheen A, Abu-Rmeileh NM, Husseini A, Abu-Raddad LJ, Khoja T, Al Rayess ZA, AlBuhairan FS, Hsairi M, Alomari MA, Ali R, Roshandel G, Terkawi AS, Hamidi S, Refaat AH, Westerman R, Kiadaliri AA, Akanda AS, Ali SD, Bacha U, Badawi A, Bazargan-Hejazi S, Faghmous IA, Fereshtehnejad SM, Fischer F, Jonas JB, Kuate Defo B, Mehari A, Omer SB, Pourmalek F, Uthman OA, Mokdad AA, Maalouf FT, Abd-Allah F, Akseer N, Arya D, Borschmann R, Brazinova A, Brugha TS, Catala-Lopez F, Degenhardt L, Ferrari A, Haro JM, Horino M, Hornberger JC, Huang H, Kieling C, Kim D, Kim Y, Knudsen AK, Mitchell PB, Patton G, Sagar R, Satpathy M, Savuon K, Seedat S, Shiue I, Skogen JC, Stein DJ, Tabb KM, Whiteford HA, Yip P, Yonemoto N, Murray CJ, Mokdad AH. The Burden of Mental Disorders in the Eastern Mediterranean Region, 1990-2013. PLoS One. 2017 Jan 17;12(1):e0169575. doi: 10.1371/journal.pone.0169575. eCollection 2017. PMID 28095477
- [Derived] Sherif Y, Fattah Azman AZ, Said SM, Siddiqah Alimuddin A, Awang H, Mohammadzadeh M. Effect of online intervention based on life skills for mental health, self-efficacy and coping skills among Arab adolescents in the Klang Valley, Malaysia: A cluster randomised controlled trial protocol. PLoS One. 2024 Feb 23;19(2):e0298627. doi: 10.1371/journal.pone.0298627. eCollection 2024. PMID 38394185